CLINICAL TRIAL: NCT00256958
Title: Static and Dynamic Balance During Standing and Walking in Correlation With Quality of Life, in Primary Total Knee Replacement
Brief Title: Static and Dynamic Balance in Correlation With Quality of Life, in Primary Total Knee Replacement
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TKR-BM-HMO-CTIL
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2005-11

CONDITIONS: Osteoarthritis; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

INTERVENTIONS:
Procedure: total knee replacement

SUMMARY:
Knee osteoarthritis (OA) is one of the most prevalent musculoskeletal complaints worldwide, affecting 30-40% of the population by the age of 65 yr.Individuals with knee OA suffer progressive loss of function.Balance is an integral component of these and many other activities of daily living. Individuals with knee OA display impairment in postural control, mostly under dynamic testing condition. Total knee replacement (TKR) has an established place in the treatment of knee osteoarthritis and is considered to be an effective intervention.It remains unknown whether TKR impact significantly at balance state of the patients with OA and whether improving in functional abilities after TKR correlates with balance control ability in this population.The purpose of this study is to determine whether TKR have any effects on relatively new postural control measures using force platform system - Balance master, in correlation with functional balance assessment.

Methods:

Participants During a year of prospective study we plan to recruit 150 participants with symptomatic OA of the knee, hospitalizing in orthopedic department of Hadassah Hospital for primary TKR. Participants will undergo evaluation just before a surgery and a year after.They will be asked to perform Balance Master measurements, ambulation and balance tests. Additional information will be collected through a questionnaire and physical examination.

DETAILED DESCRIPTION:
Balance Master Testing

The Pro Balance Master system with software version 8 will be used in the study. The Pro Balance Master system is comprised of two 23cm × 46cm dual force plates connected at the midline of the anterioposterior axis by a pin joint. Each force plate is mounted on a pair of symmetrically positioned force transducers. The four transducers measure vertical ground reaction forces, which form the basis of subsequent calculations of center of pressure (COP) and center of gravity (COG) sway angels. All test data are acquired and then stored on a PC.

Subjects are instructed to remove their shoes and step onto the forceplates, which have to be covered with tracing paper. Their feet are positioned by aligning the lateral border of the foot with the appropriate height line marked on the forceplates (ie, short, 76 to 140 cm; medium, 141 to 165cm; or tail, 166 to 203cm). The medial maileoli are aligned with the transverse forceplate line and subjects adopted a comfortable amount of forefoot splay. The outline of their feet is traced onto paper to ensure the same placement in subsequent testing sessions. The visual display monitor is adjusted to the subject's eye level. Subjects are instructed not to move their feet and are asked to stand with their arms at their sides throughout the testing procedure. The standard test suite protocol will be administered, consisting of 6 tests, 3 of which are static and 3 dynamic. The static tests require the subject to look straight ahead while standing as still as possible, initially with eyes open, then with eyes closed, and finally focusing on the display monitor using visual feedback to maintain the position of a cursor (representing the subject's COG) within a centrally positioned target box. For each test, data relating to postural sway is recorded for a period of 20 seconds and the area of the sway is calculated and expressed as a percentage of the subject's theoretical limits of stability (LOS). Assuming that movement about the ankle (with a fixed foot position) resembles an inverted pendulum, these limits are defined as extending 6.25 ° anteriorly, 4.45 ° posteriorly, and 8.00 ° to each side, ~2 and delimit the area over which the COG can safely move without changing the base of support.

All three dynamic tests require subjects to shift their COG. The first dynamic test involves rhythmic weight shifting side to side to 50% of the LOS at 3-second then 2-second pacing. Subjects are instructed to match the timing and movement of a bail on the screen by shifting their body weight side to side to target lines denoted on the screen. The second test is similar to the first except movement was now in an anterioposterior direction. Data reflecting the average magnitude of the movement path (expressed as a percentage of the LOS) are produced from six trials at each pace for each movement direction. The absolute error relative to the targets (set at 50% of the LOS) is calculated by subtracting 50 from the score obtained (50% indicating perfect execution) and recording it in absolute terms.

The final dynamic test involved weight shifting to 8 targets positioned in an ellipse, the perimeter of which corresponded to 75% of the LOS. The subjects are required to follow a ball to each target as it is highlighted, and remain at that target for 3 seconds before returning to the central target (neutral).

Targets are highlighted in random order, but each target is selected only once. The maximum allowable movement time to reach a target is 8 seconds. The average movement time and path sway (in terms of percentage of the LOS) is determined across targets. A score of 100% indicated that no path deviation had occurred, ie, perfect execution. (It should be noted that the processing of the data to produce the outcome measures described above is hard coded by NeuroCom.ª)

Main Outcome Measures:

Oxford Knee Score (OKS). The OKS is a self-completed patient based outcome score . It is a 12 item self-completed patient based outcome score. The questionnaire was developed from patient interview and validated against two generic health scales, the SF-36 and Health Assessment Questionnaire (HAQ) [44]. It was originally intended for use in large randomised controlled trials for patients undergoing total knee replacement, to assess levels of, and changes in, pain and function of the knee solely from the patient's viewpoint. Data collection can be via a postal questionnaire or by directed interview.

Visual Analog Scale (VAS).The severity of knee pain is evaluated by the VAS [45] after patients remain in a weight-bearing position (walking or standing) for 5 minutes in the parallel bars. The VAS instrument consisted of horizontal lines 10cm long, with anchor points of 0 (no pain) and 10 (maximum pain).

Four Square Step Test (FSST). FSST is a clinical measure of rapid stepping and obstacle avoidance . The equipment required for the FSST includes a stopwatch and 4 canes. The square is formed by using 4 canes resting flat on the floor. Canes are 90cm long, and the direction and type of handle used is not important. The subject stands in square number 1 facing square number 2. The aim is to step as fast as possible into each square in the following sequence. Square number 2, 3, 4, 1, 4, 3, 2, and 1. This sequence requires the subject to step forward, backward, and sideway to the right and left. The score is recorded as the time taken to complete the sequence. The stopwatch starts when the first foot contacts the floor in square 2 and finishes when the last foot comes back to touch the floor in square 1. The following instructions are given to the subject, "Try to complete the sequence as fast as possible without touching the sticks. Both feet must make contact with the floor in each square. If possible, face forward during the entire sequence." The sequence is then shown to the subject.

One practice trial is completed to ensure the subject knows the sequence. Two FSST are completed with the best time taken as the score. A trial is repeated if the subject fails to complete the sequence successfully, loses balance, or makes contact with a cane during the sequence. Subjects who were unable to face forward during the entire sequence and needed to turn before stepping into the next square were still given a score. All subjects wore their preferred shoes. The examiner stood in a position to see all steps taken by the subject, and an assistant provided the subject with close supervision. The entire test, including giving instructions and a practice trial, took less than 5 minutes to complete.

Time Up and Go test (TUG). Subjects are required to stand up from a chair with armrests, walk 3m, turn around, return to the chair, and sit down. The time taken to complete this task is measured in seconds with a stopwatch [47]. The TUG test showed a high degree of test-retest reliability in TUG scores in elderly subjects .

SF-36. This is a 36-item questionnaire which measures health functioning on eight scales, including a physical functioning scale, and is among the most widely used measures of quality of life in studies of patients and populations .Missing data and scoring procedures followed the SF-36 user guidelines .

ELIGIBILITY:
Inclusion Criteria:During a year of prospective study we plan to recruit 150 participants with symptomatic OA of the knee, hospitalizing in orthopedic department of Hadassah Hospital for primary TKR. Confirmation of diagnosis of OA will be based on the American College of Rheumatology classification criteria . Participants have to be able to stand and to walk and also to follow simple instructions.

-

Exclusion Criteria:previous knee surgery, neurological problem with severe motor deficit (Parkinson disease, hemiplegia, spinal cord injury), severe orthopedic problem of low limbs (arthrodesis of low limb's joints, failed TKR/THR, amputation, failed back), systemic arthritic condition, severe cognitive problem with restricted consent.

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-11; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Balance Master Testing
Oxford Knee Score
Visual Analog Scale
Four Square Step Test
Time Up and Go test

SECONDARY OUTCOMES:
SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Schwartz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel